CLINICAL TRIAL: NCT00118443
Title: RCT of Gatekeeper Training for Suicide Prevention
Brief Title: Evaluation of a School-Based Training Program for Suicide Prevention
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Peter Wyman, PhD, University of Rochester Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34MH071189 (NIH); R34MH071189 (NIH); DSIR 82-SEDR
Record Dates: First submitted 2005-07-06; First posted 2005-07-11 (Estimated); Last update posted 2013-06-28 (Estimated); Status verified 2013-06

CONDITIONS: Suicide
Keywords: Suicide Prevention; Depression; Adolescent; Students; School Teachers
MeSH Terms: conditions — Suicide; Suicide Prevention; Depression | interventions — Referral and Consultation

INTERVENTIONS:
Behavioral: Question, Persuade, Refer (QPR) training

SUMMARY:
This study will determine whether a training program designed to help school staff members identify adolescents at risk for suicide will increase the number of students who are referred to mental health services.

DETAILED DESCRIPTION:
The rate of suicide among adolescents has significantly increased in recent years. Psychiatric disorders are often associated with increased suicide risk; therefore, the ability to identify adolescents with signs of depression and other psychiatric conditions is clear. This study will determine the effectiveness of a suicide prevention training program called Question, Persuade, Refer (QPR) in increasing the number of potentially suicidal adolescents who are referred to mental health services. The training is designed to help school staff recognize signs that a student may be suicidal, provide tips on how to question students about any suicidal thoughts they may have, and provide techniques to persuade students to seek suicide prevention help.

School staff will be randomly assigned to either receive QPR training for 2 years starting immediately or be placed on a waiting list for later training. The rates of referral to the school district's prevention/intervention centers will be used to assess the effectiveness of QPR training. In addition, the impact of QPR training on school staff members' knowledge and attitudes about intervening with at-risk students will be assessed through surveys at four time points over the 2-year study duration with a randomly selected portion of staff in the 32 participating schools. Surveys completed by randomly selected 8th and 10th grade students will also be used to determine whether the intervention is effective in reducing suicidal thoughts or attempts.

Study hypothesis: More students in schools that have Question, Persuade, Refer (QPR)-trained staff will be referred for a mental health evaluation than in schools without QPR-trained staff.

ELIGIBILITY:
Inclusion Criteria for School Staff Members:

* Currently working as a staff member in Cobb County school district

Inclusion Criteria for Students:

* Parent or guardian willing to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 50000 (Estimated)
Dates: Start 2004-03; Primary Completion 2006-12 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Rates of referrals for students identified as suicidal risks
school staff knowledge and attitudes
outcomes of mental health evaluations for accurate detection of suicidal risk

CONTACTS AND LOCATIONS:
Overall Officials: Peter Wyman, PhD, Principal Investigator — University of Rochester
Locations (1):
- Cobb County School District, Marietta, Georgia, United States